CLINICAL TRIAL: NCT05756816
Title: SurePulse Oximeter - a Targeted Oxygenation Observation: A Controlled Desaturation Study to Establish the Accuracy and Precision of the SurePulse VS Patch Newborn Vital Sign Monitor (VSP)
Brief Title: SurePulse Oximeter - a Targeted Oxygenation Observation
Acronym: SPO-TOO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Surepulse Medical Limited (Industry)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VSP-CI-01; MTT-ISG-INS-196 (Other Grant/Funding Number: Medilink East Midlands); 317814 (Other: IRAS)
Record Dates: First submitted 2023-02-03; First posted 2023-03-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Hypoxia; Oxygen Saturation; Pulse Oximetry
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: A controlled and stepwise reduction in oxygen blood levels, with both the SurePulse VS and SurePulse VSP placed on the volunteer.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SurePulse VS and VSP devices (Experimental): All enrolled participants will undergo a controlled and stepwise reduction in oxygen blood levels, with both the SurePulse VS/SurePulse VSP placed on the volunteer.
  Interventions: Device: SurePulse VSP; Device: SurePulse VS

INTERVENTIONS:
Device: SurePulse VSP — A controlled and stepwise reduction in oxygen blood levels in healthy volunteers, with the SurePulse VSP placed on the volunteer.
Device: SurePulse VS — A controlled and stepwise reduction in oxygen blood levels in healthy volunteers, with the SurePulse VS placed on the volunteer.

SUMMARY:
This clinical investigation will investigate how accurate the SurePulse VS and SurePulse VS Patch (VSP) are for measuring blood oxygen levels (oxygen saturation). If the results are accurate, the VSP will be ready to apply for regulatory approval, meaning it could then be available for use on newborn babies in the National Health Service (NHS).

DETAILED DESCRIPTION:
Healthy volunteers who express an interest in the study and meet the eligibility criteria will be invited to participate in the study. This study will investigate the accuracy and safety of the SurePulse VS and SurePulse VS Patch (VSP) in measuring blood oxygen levels. This is done by measuring blood oxygen levels across a range of values in healthy adults. The measurements from the VS and VSP will be compared to the known correct value. The study follows the internationally agreed standard for pulse oximeter approval.

Agreeing participants will have their name, contact details, medical history, height, weight, date of birth, skin colour, emergency contact details and address recorded, as necessary to conduct the study. After completion of the eligibility and consent process, participants will be enrolled in the study. Healthy volunteers will have their blood oxygen levels temporarily reduced in a controlled and stepwise manner. Oxygen levels will not be low for the entire duration of the session. Oxygen levels will be reduced to a specific target for a few minutes at a time. Volunteers will have a small tube inserted into an artery (blood vessel) in their wrist; this will be used to take blood samples throughout the session. The blood samples will be taken, analysed and destroyed in the same room. The session should take approximately 1.5 - 2 hours in total.

The output from the study will be compared to the primary and secondary outcomes to evaluate the performance and safety of the device. This study is required for the SurePulse VSP to be regulatory approved, meaning it could then become available in the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55
* Willing and able to provide written informed consent
* Healthy adult subjects (ASA 1)
* Non-smoker
* Willing and able to comply with study procedures and duration

Exclusion Criteria:

* Smokers or individuals exposed to high levels of carbon monoxide
* Compromised circulation, injury, or physical malfunction of the sensor sites which would limit the ability to test sites needed for the study
* Female subjects that are actively trying to get pregnant or are pregnant (conﬁrmed by Health Assessment Form). N.B. All female participants will be offered a pregnancy test
* Unwillingness or inability to remove coloured nail polish from test digits (relevant for reference pulse oximeter) or to have medical monitoring attached
* Known health conditions disclosed on Health Assessment Form which mean that participant is not healthy
* Allergy to lidocaine
* Allergy to adhesives used in medical dressings or tapes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — There should be a minimum of 40% male and minimum of 40% female participants with the balance made up of either.
Enrollment: 19 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Validation of the SpO2 accuracy of the SurePulse VS Patch Newborn Vital Sign Monitor (VSP) pulse oximeter in comparison to "gold-standard" measurements of blood SaO2 by a co-oximeter. | Through study completion, an average of 2 hours
  Oxygen saturation comparison of measurements taken by the SurePulse VSP (SpO2) and co-oximeter blood gas analyser (SaO2). For the statistical analysis, the Accuracy Root Mean Square (Arms) calculation is used to determine the SpO2 accuracy performance.
Adverse events (AEs) attributable to the SurePulse medical devices | Through study completion, an average of 2 hours
  Incidence, severity and causality of all AEs with delineation of those that are attributable to the use of the SurePulse medical devices to be used as a measure of device safety. Safety is measured by adverse events attributable to SurePulse medical devices and will be measured by adverse event logs and reports and their associated reporting requirements.

SECONDARY OUTCOMES:
Validation of the SpO2 accuracy of the SurePulse VS Monitor (VS) in comparison to "gold-standard" measurements of blood SaO2 by a co-oximeter. | Through study completion, an average of 2 hours
  Oxygen saturation comparison of measurements taken by the SurePulse VS (SpO2) and co-oximeter blood gas analyser (SaO2). For the statistical analysis, the Accuracy Root Mean Square (Arms) calculation is used to determine the SpO2 accuracy performance.
Validation of the pulse rate accuracy of the SurePulse VS Patch Newborn Vital Sign Monitor (VSP) pulse oximeter in comparison to ECG. | Through study completion, an average of 2 hours
  Pulse Rate comparison of measurements taken by the SurePulse VSP and ECG. For the statistical analysis, the Accuracy Root Mean Square (Arms) calculation is used to determine the Pulse Rate accuracy performance.
Validation of the pulse rate accuracy of the SurePulse VS Monitor (VS) in comparison to ECG. | Through study completion, an average of 2 hours
  Pulse Rate comparison of measurements taken by the SurePulse VS and ECG. For the statistical analysis, the Accuracy Root Mean Square (Arms) calculation is used to determine the Pulse Rate accuracy performance.

CONTACTS AND LOCATIONS:
Overall Officials: Murray du Plessis, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No